CLINICAL TRIAL: NCT06625346
Title: Clinical Outcomes in Newly Diagnosed Hypertensive Patients With EXTOR (Fixed-Dose Combination of Amlodipine/Valsartan) in Routine Pakistani Practice.
Brief Title: Clinical Response of EXTOR (Amlodipine/Valsartan) in Newly Diagnosed Hypertensive Patients.
Acronym: HELP
Status: Recruiting | Type: Observational
Sponsor: The Searle Company Limited Pakistan (Industry)
Responsible Party: Sponsor
Other Study IDs: TSCL-HELP-01
Record Dates: First submitted 2024-03-19; First posted 2024-10-03 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
Keywords: Hypertnsion; Amlodipine valsartan combination; Quality of life (QoL); Pakistan
MeSH Terms: conditions — Hypertension | interventions — Valsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Naive Hypertensive patients: Naive Pakistani subjects diagnosed as the case of Hypertension prescribed Extor in routine practice.
  Interventions: Drug: Fixed-Dose Combination of Amlodipine/Valsartan

INTERVENTIONS:
Drug: Fixed-Dose Combination of Amlodipine/Valsartan — Amlodipine and valsartan are two of the most commonly prescribed medications for the treatment of hypertension (high blood pressure). Amlodipine is a calcium channel blocker that works by relaxing the blood vessels, while valsartan is an angiotensin receptor blocker that works by blocking the effects of the hormone angiotensin II, which causes blood vessels to constrict. The combination of amlodipine and valsartan in a single pill has been shown to be more effective in lowering blood pressure than either medication alone. This is because the two medications have different mechanisms of action and work together to provide a more comprehensive approach to blood pressure control.
  Other Names: EXTOR

SUMMARY:
The American College of Cardiology/American Heart Association hypertension guidelines recommend treatment initiation with dual antihypertensive therapy in adults with stage 2 hypertension (corresponding to grade 1 and 2 in the ESH classification) and an average BP >20/10 mm Hg above target. Amlodipine and valsartan are two of the most commonly prescribed medications for the treatment of hypertension (high blood pressure). In Pakistan multiple studies were conducted on Hypertension and use of Single Pill Combination in uncontrolled Hypertension. However, no study was conducted to assess the role of Single Pill Combination (SPC) like Amlodipine and Valsartan in newly diagnosed hypertension and to assess their quality of life by patients' satisfaction with their medication after managing the hypertension with the SPC.

DETAILED DESCRIPTION:
To assess the effectiveness of EXTOR (Amlodipine/Valsartan) in newly diagnosed hypertensive patients in 8 weeks.

* Change from Baseline to 8 weeks in Systolic Blood Pressure (SBP) From standard Blood Pressure Measurement.
* Change from Baseline to 8 weeks in Diastolic Blood Pressure (DBP) From standard Blood Pressure Measurement.
* Change from Baseline to 8 weeks in the Health-Related Quality of Life of newly diagnosed hypertensive patients managed by Extor: assess by Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9)
* Change from baseline to 4 weeks in Diastolic Blood Pressure (SBP) From standard Blood Pressure Measurement
* Change from baseline to 4 weeks in Diastolic Blood Pressure (DBP) From standard Blood Pressure Measurement
* Change from baseline to 4 weeks in the Health-Related Quality of Life of newly diagnosed hypertensive patients managed by Extor: assess by Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9)
* To assess the overall safety of EXTOR (Amlodipine/Valsartan) in newly diagnosed hypertensive patients.

Note: The safety is assessed in all subjects who received at least one dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a clinical history of Hypertension (systolic blood pressure greater than or equal to 140 mmHg or a diastolic blood pressure greater than or equal to 90 mmHg) and never had antihypertensive treatment.
* Patient aged ≥18 and ≤70 years inclusive of either sex.
* Patient with ability to understand and sign written informed consent form.

Exclusion Criteria:

* • Patients with already on antihypertensive treatment or secondary hypertension

  * Pregnant women or nursing mothers
  * Patients with acute illnesses or psychiatric diagnosis
  * Known hypersensitivity to Extor product, the metabolites, or formulation excipients.
  * Treated with Extor to evaluate safety as per approved prescribing information for Extor in Pakistan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will be enrolled as per inclusion/exclusion criteria in the study. The total sample size of the study is 420 subjects with Hypertension for the multiple selected study sites and this will have 95% power to detect mean change from baseline to week 4-and 8 weeks for the evaluation of the effectiveness and overall safety response of Extorl for the Essential Hypertension treatment, assuming a standard deviation of the differences of 15.5, using 0.05 two-sided significance level considering 10% drop-out rate
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of EXTOR (Amlodipine/Valsartan) in newly diagnosed hypertensive patients in 8 weeks. | 8 week
  * Change from Baseline to 4 week and 8 weeks in Systolic Blood Pressure (SBP) From standard Blood Pressure Measurement. The achieve BP control defined as systolic BP less than 140 mmHg at any of their clinic visits and maintained at the 8 week of treatment clinic visit.
  * Change from Baseline to 4 week and 8 weeks in Diastolic Blood Pressure (DBP) From standard Blood Pressure Measurement. The achieve BP control defined as Diastolic BP less than 90 mmHg at any of their clinic visits and maintained at the 8 week of treatment clinic visit.
To assess the Health-Related Quality of Life of newly diagnosed hypertensive patients managed by Extor | 8 week
  • Change from Baseline to 4 week and 8 weeks in the Health-Related Quality of Life of newly diagnosed hypertensive patients managed by Extor, assess by Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9). For TSQM-9 questionnaire applies to assesses patient satisfaction with Extor medication including Effectiveness (3 items), Convenience (2 items), Side effects (2 items) and Global satisfaction (2 items). The TSQM-9 score from 01 to 07. The 01 score (minimum) is Extremely Dissatisfied and Score 07 (maximum) is Extremely Satisfied
To assess the overall safety of EXTOR (Amlodipine/Valsartan) in newly diagnosed hypertensive patients. | 8 week
  Safety & tolerability will assess based on the incidence of reported TEAEs by system organ class ; preferred term, as well as by categories: TEAE, severe TEAE, serious TEAE, drug-related TEAE, drug-related severe TEAE, drug-related serious TEAE, TEAE leading to discontinuation, & TEAE with outcome of death. Drug-related TEAEs were defined as TEAEs assigned a Study Drug (Extor) relationship of adverse reaction & suspected adverse reaction.
  TEAEs were coded using the Medical Dictionary for Regulatory Activities, version 19.0. The severity of TEAEs are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03. TEAEs were defined as any adverse event that started or increased in severity after the first dose of Study Drug on Day 1 through the Final Study Visit (8 weeks +/-3 days after last dose).

CONTACTS AND LOCATIONS:
Overall Officials: Asif Mahmood, MBBS, MPH, Study Director — The Searle Company Limited Pakistan
Locations (2):
- Pakistan (2):
  - Kuwait Teaching Hospital, Peshawar, KPK
  - National Medical Centre, Karachi

IPD SHARING:
Plan to Share IPD: No